CLINICAL TRIAL: NCT03547609
Title: Study on the Mnemic Functioning of Children With Kabuki Syndrome
Brief Title: Assessment of Memory in Children With Kabuki Syndrom
Acronym: MEM-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5005
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-05

CONDITIONS: Kabuki Syndrome
Keywords: Kabuki Syndrome; Intellectual Profile; Memory
MeSH Terms: conditions — Kabuki syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No arm intervention — No arm intervention

SUMMARY:
Mnesic function has not, at present, been evaluated in patients with Kabuki Syndrome. Some data from the neuroimagery suggest an impairment of memory function. The objective of our study is to assess the mnesic function of children with Kabuki Syndrom.

DETAILED DESCRIPTION:
Kabuki Syndrome (SK - OMIM 147920 and 300867 ORPHA: 2322) is a rare genetic disease with a prevalence of approximately 1/32 000 and responsible for a malformation syndrome with mild to moderate intellectual impairment. SK is due to mutations in the KMT2D and KDM6A genes. As part of a national PHRC (AOM 07-090, clinicaltrial NCT01314534, The investigators were able to perform psychometric tests type WISC4 and MRI type VBM). Disability in SK is characterized by a heterogeneous cognitive profile with strengths and weaknesses when calculating IQ. Brain MRI reveals small hippocampi compared to controls. These 2 data are partly contradictory because the strengths of the patients with SK are a working memory and a verbal comprehension index high compared to the other indices of the tests WISC-IV.

The objective of the research is to better understand the mnesic function of children with SK.

25 children aged 6 to 16 will be recruited. The diagnosis of SK will have been authenticated by the demonstration of a mutation in the KMT2D or KDM6A gene.

The memory assessments will be conducted in one visit for each child, who will perform a memory assessment with a neuropsychologist, using the CMS scale.

ELIGIBILITY:
Inclusion Criteria:

* Child from 6 to 16 years old
* Presents an already established diagnosis of Kabuki syndrome.
* Free, informed and written consent signed by the participant's parents, and the investigator (at the latest inclusion day and before any research required by the research).

Exclusion Criteria:

* Be under 6 years old or over 16 years old
* Do not master the French language
* Not having access to language
* Deafness not paired
* Blindness.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
CMS (selective motor control scale) main score | 1 hour
  CMS main score

SECONDARY OUTCOMES:
CMS (selective motor control scale) indexes | 1 hour
  CMS indexes

CONTACTS AND LOCATIONS:
Locations (1):
- Genetic Departement, rare disease, personalized medicine, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lehman N, Mazery AC, Visier A, Baumann C, Lachesnais D, Capri Y, Toutain A, Odent S, Mikaty M, Goizet C, Taupiac E, Jacquemont ML, Sanchez E, Schaefer E, Gatinois V, Faivre L, Minot D, Kayirangwa H, Sang KLQ, Boddaert N, Bayard S, Lacombe D, Moutton S, Touitou I, Rio M, Amiel J, Lyonnet S, Sanlaville D, Picot MC, Genevieve D. Molecular, clinical and neuropsychological study in 31 patients with Kabuki syndrome and KMT2D mutations. Clin Genet. 2017 Sep;92(3):298-305. doi: 10.1111/cge.13010. Epub 2017 May 18. PMID 28295206